CLINICAL TRIAL: NCT06019650
Title: Elderly Culturally Adapted Manual Assisted Brief Psychological Therapy (E-CMAP) for Older Adults With Suicidal Ideation: An Exploratory Randomized Controlled Trial From Pakistan
Brief Title: Culturally Adapted Suicide Prevention Intervention for Older Adults
Acronym: ECMAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ECMAP
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Suicidal Ideation
Keywords: suicidal ideation,; self-harm; older adult; elderly; ECMAP; Pakistan; LMIC
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-CMAP Intervention (Experimental): CMAP is a culturally adapted brief problem-focused therapy, based on the principles of CBT which has been adapted with permission from a self-help guide called "Life after self-harm"(Schmidt & Davidson, 2004). This intervention includes evaluation of the self-harm attempt, crisis skills, problem-solving and basic cognitive techniques to manage emotions, negative thinking and relapse prevention strategies.
  Interventions: Behavioral: ECMAP
- Standard Routine Care (No Intervention): Local medical, psychiatric and primary care services provide standard routine care according to their clinical judgment and available resources

INTERVENTIONS:
Behavioral: ECMAP — The therapist will deliver 12-week training program comprised of 6 sessions at the participant's home/outpatient clinic depending upon the participants' choice within 3 months. The first two sessions will be offered weekly and then fortnightly.
  Arms: E-CMAP Intervention

SUMMARY:
determine the efficacy of culturally adapted manual assisted brief psychological intervention for older adults (E-CMAP) with suicidal ideation

DETAILED DESCRIPTION:
Suicide is a serious public health concern. Each year more than 800,000 people worldwide die due to suicide. Most of these (79%) are in the low and middle-income countries (LMIC), with an increased risk of suicide in ageing.

Primary Objective: To assess the effectiveness of E-CMAP compared to Treatment as Usual (TAU) as measured by reduction in suicidal ideation third month post-randomization with Beck Scale for Suicidal ideation (BSI) (Beck & Steer, 1991) Secondary outcomes: the two groups will be compared on hopelessness, depression, quality of life, coping skills, participant satisfaction, health/social care usage, and episodes of self-harm. All variables known to be related to suicide risk.

The study will be carried out in two stages. First stage will be cultural adaptation and refinement of the intervention and second stage will be feasibility Randomised Control Trial (RCT).

Stage 1: In the first stage, the adaptation of the intervention for suicidal ideation in older adults will be carried out by a group of experts including a master trainer, a bilingual health expert, mental health professional potential user (i.e., older adults with suicidal ideation), and a senior therapist through discussion groups.

Stage 2: Feasibility randomized controlled trial (RCT) After adaptation, the intervention will be tested in a multicenter RCT to determine the efficacy of culturally adapted manual assisted brief psychological intervention for older adults/elderly (E-CMAP) with suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

In the context of this study, suicidal ideation is defined as; "Passive thoughts about wanting to be dead or active thoughts about killing oneself, these thoughts may include plan but not accompanied by preparatory behavior" (Griffin et al., 2020)

* 50 years and above
* Has recent history of experiencing suicidal ideation
* Participants living within the catchment area of the participating practices and hospitals.
* Capacity to give informed consent.

Exclusion Criteria:

* Unable to provide consent due to severe mental or physical illness.
* Unlikely to be available for outcome assessments (temporary residence)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | change in total scores from baseline to 3-month post randomization assessment
  Participants suicidal ideation will be assessed using the Beck scale for suicidal ideation. Higher scores on the questionnaire indicate greater severity of suicidal ideation. Scores provide a measure of the severity of self-reported hopelessness: 0-3 minimal, 4-8 mild, 9-14 moderate, and 15-20 severe.

SECONDARY OUTCOMES:
Hopelessness | change in total scores from baseline to 3-month post randomization assessment
  Participants feelings of hopelessness will be assessed using the Beck Hopelessness Scale. Higher scores indicate greater severity of hopelessness. Scores ranging from: 0 to 3 as are considered within the normal range, 4 to 8 identify mild hopelessness, scores from 9 to 14 identify moderate hopelessness, and scores greater than 14 identify severe hopelessness
Depression | change in total scores from baseline to 3-month post randomization assessment
  Participants severity of depression will be assessed using the Beck Depression Inventory. Higher scores indicate greater severity of depression. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Health-related Quality of Life | change in total scores from baseline to 3-month post randomization assessment
  Participants Health related quality of life will be assessed using the EQ-5D- 5L. Higher scores indicate better health related quality of life
Coping Resource Inventory | change in total scores from baseline to 3-month post randomization assessment
  Participants coping skills will be assessed using the Coping Resource Inventory. Higher scored indicate better coping skills.
Client Satisfaction Questionaire | level of satisfaction at end of intervention i.e., 3-month post-randomization
  Participant satisfaction with services will be assessed using the Client Satisfaction Questionnaire. Higher scores indicate greater level of satisfaction with the services.
Service Usage | change in total scores from baseline to 3-month post randomization assessment
  Service usage (including formal (GPs/ other doctor and informal sector such as faith healers/imams) will be assessed using client service receipt inventory. There are no score ranges for this scale.
Episodes of Self-harm | change in total scores from baseline to 3-month post randomization assessment
  Episodes of Self-harm will be assessed using the Suicide attempt self -injury interview. This is the semi-structured instrument to assess different aspects of episode of self-harm. This scale does not have any cut-off or score ranges.
Problem Solving Skills | change in total scores from baseline to 3-month post randomization assessment
  Participants problem Solving skills will be assessed using Problem solving Inventory. Higher scores indicate better problem solving skills. The possible total scale score of PSI ranges between 32 and 192.

CONTACTS AND LOCATIONS:
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husain N, Kiran T, Chaudhry IB, Williams C, Emsley R, Arshad U, Ansari MA, Bassett P, Bee P, Bhatia MR, Chew-Graham C, Husain MO, Irfan M, Khaliq A, Minhas FA, Naeem F, Naqvi H, Nizami AT, Noureen A, Panagioti M, Rasool G, Saeed S, Bukhari SQ, Tofique S, Zadeh ZF, Zafar SN, Chaudhry N. A culturally adapted manual-assisted problem-solving intervention (CMAP) for adults with a history of self-harm: a multi-centre randomised controlled trial. BMC Med. 2023 Jul 31;21(1):282. doi: 10.1186/s12916-023-02983-8. PMID 37525207